CLINICAL TRIAL: NCT01339286
Title: Study of Associated Gene Polymorphisms With Atomoxetine Response Prediction in ADHD Treatment
Brief Title: Associated Genes With Atomoxetine Response in Attention Deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Li Yang, Peking University the Sixth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSFC30800302
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- atomoxetine (Experimental)
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: atomoxetine — Atomoxetine will be titrated to optimal dose, beginning with 0.5mg/kg.d, then increasing to 1.2mg/kg.d in two weeks and maintaining for 4 weeks. If the optimal dose does not achieved, the dose can be increased further to 1.4mg/kg.d and maintained for 4 weeks.

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is the most common behavior disorder, with the prevalence of 3% to 6% in children and adolescents. The patients' academic achievements, professions and social livings are impaired. Comorbid antisocial behavior, substance abuse and delinquency burden family and society. Stimulants used to be the first line drug. But the medication compliance is poor because of strict drug administration. Atomoxetine is a new non-stimulant drug, which can effectively improve ADHD symptoms. But it achieves effect slowly, the drug responses differ significantly, and side effects interfere compliance. Since genetic factors is the most important cause for different drug responses, this project studies candidate genes potentially associated with atomoxetine medication, with the aim to find 2 to 3 gene polymorphisms influencing the drug response of ADHD. The study adopts cohort design. A sample of more than 100 ADHD cases with atomoxetine medication is to be collected. The rapid genotyping of large sample depends on high-through laboratory. New statistic method is to be used to improve the sensitivity of the target gene detection. There has been no such report in country and overseas. This project will provide basic information for forecasting drug response, improving clinical effects, tolerance and long-term compliance.

ELIGIBILITY:
Inclusion Criteria:

* The subject should meet with the DSM-IV ADHD criteria, confirmed by semi-structured interview.
* The subject has not accepted any treatment for ADHD before, or he/she received methylphenidate or atomoxetine treatment but has stopped for 1 or 4 weeks respectively.
* Han Chinese
* Parent sign the informed consent

Exclusion Criteria:

* Who are allergy to atomoxetine
* Who can not complete the titration procedure because of untolerable of the side effect
* Who combined other psychotropic drugs or non-drug intervention for ADHD.
* Children who can not be compliant with the blood withdraw.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of ADHD symptoms as rated by ADHD Rating Scale: IV (Investigator Rated) | an expected average of 8 weeks
  Change from baseline in ADHD Rating Scale: IV (Investigator Rated) after optimal dose treated for 4 weeks

SECONDARY OUTCOMES:
Improvement of ADHD symptoms as rated by ADHD Rating Scale: IV (Parent Rated) | an expected average of 8 weeks
  Change from baseline in ADHD Rating Scale: IV (Parent Rated) after optimal dose treated for 4 weeks
Improvement of ADHD symptoms as rated by ADHD Rating Scale: IV (Teacher Rated) | An expected average of 8 weeks
  Change from baseline in ADHD Rating Scale: IV (Teacher Rated) after optimal dose treated for 4 weeks
Improvement of behaviors as rated by IOWA Conners Rating Scale (Parent Rated) | An expected average of 8 weeks
  Change from baseline in IOWA Conners Rating Scale (Parent Rated) after optimal dose treated for 4 weeks
Improvement of behaviors as rated by IOWA Conners Rating Scale (Teacher Rated) | An expected average of 8 weeks
  Change from baseline in IOWA Conners Rating Scale (Teacher Rated) after optimal dose treated for 4 weeks
Improvement in Clinical Global Impression: Severity | An expected average of 8 weeks
  Change from baseline in Clinical Global Impression: Severity after optimal dose treated for 4 weeks
Side effect | An expected average of 8 weeks
  Number of Subjects with Side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China